CLINICAL TRIAL: NCT04310761
Title: Retrospective Comparison of Pregnancy Outcome of Infertile Patients After Fresh and Warmed Single Blastocyst Transfer From 2014 to 2018.
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: XX/2020
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Primary Maternal and Neonatal Outcomes; Assisted Reproductive Technology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pregnancy population after one single blastocyst transfer: The data have been collected from the Humanitas Fertility Center' Department database (ART.it) from a period between 2014 and 2018.
  Interventions: Procedure: one single blastocyst transfer, both fresh and warmed

INTERVENTIONS:
Procedure: one single blastocyst transfer, both fresh and warmed — Ultrasound guided transvaginal embryo transfer.

SUMMARY:
The investigators retrospectively analysed the maternal and neonatal outcomes following a single fresh blastocyst transfer and a single warmed blastocyst transfer from procedures performed between 2014 and 2018 in a tertiary level university based fertility clinic.

DETAILED DESCRIPTION:
Previous studies that analysed pregnancy outcomes in women who underwent frozen single blastocyst transfer have shown an increase rate of large for gestational age and very large for gestational age (Zhang et al., 2019),increased maternal risks of placenta accreta and pregnancy-induced hypertension (Ishihara et al.,2014),and lower risks of placenta previa, placental abruption, very pre-term birth, small for gestational age, and perinatal mortality (Sha, Yin, Cheng,& Massey, 2018) than fresh blastocyst transfer.

The main outcome of this study is to analyse the rate of live births with the relative gestational period and neonatal weight and still death and neonatal death per each single blastocyst transfer, both fresh and warmed. Secondary outcomes include the incidence of obstetric pathologies, gestational diabetes and pre-eclampsia, and defects of placentation.

The study database included all pregnancies occurred after both a single fresh and warmed blastocyst transfer between the five-year period from 2014 to 2018 at Humanitas Fertility Centre. The inclusion criteria were all patients, without any age limitations, which underwent either FIVET or ICSI and only transferred a single blastocyst. With regards to exclusion criteria, the following were considered: ovodonation, suspended cycles and embryos which were subjected to pre-implantation genetic testing.The investigator performed a comparison of maternal and neonatal outcomes in these pregnancies which occurred in the same period of time and in the same age-group of women.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women, without any age limitations, which underwent either FIVET or ICSI and only transferred a single blastocyst (warmed or fresh).

Exclusion Criteria:

* Ovodonation, suspended cycles, and embryos subjected to pre-implantation genetic testing.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All infertile patients which performed a single fresh and a single frozen embryo transfer from 2014 to 2018.
Sampling Method: Probability Sample
Enrollment: 4613 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of live births | 5 years
  Rate of live births with the relative gestational period and neonatal weight and still death and neonatal death per each single blastocyst transfer, both fresh and warmed

SECONDARY OUTCOMES:
Incidence of obstetric pathologies | 5 years
  Incidence of obstetric pathologies, gestational diabetes and pre-eclampsia, and defects of placentation.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang J, Wang Y, Liu H, Mao X, Chen Q, Fan Y, Xiao Y, Kuang Y. Effect of in vitro culture period on birth weight after vitrified-warmed transfer cycles: analysis of 4,201 singleton newborns. Fertil Steril. 2019 Jan;111(1):97-104. doi: 10.1016/j.fertnstert.2018.10.006. Epub 2018 Nov 17. PMID 30458993
- [Background] Ishihara O, Araki R, Kuwahara A, Itakura A, Saito H, Adamson GD. Impact of frozen-thawed single-blastocyst transfer on maternal and neonatal outcome: an analysis of 277,042 single-embryo transfer cycles from 2008 to 2010 in Japan. Fertil Steril. 2014 Jan;101(1):128-33. doi: 10.1016/j.fertnstert.2013.09.025. Epub 2013 Oct 23. PMID 24268706
- [Background] Sha T, Yin X, Cheng W, Massey IY. Pregnancy-related complications and perinatal outcomes resulting from transfer of cryopreserved versus fresh embryos in vitro fertilization: a meta-analysis. Fertil Steril. 2018 Feb;109(2):330-342.e9. doi: 10.1016/j.fertnstert.2017.10.019. Epub 2018 Jan 11. PMID 29331236
- [Derived] Cirillo F, Grilli L, Ronchetti C, Paladino I, Morenghi E, Busnelli A, Levi-Setti PE. Retrospective comparison of pregnancy outcomes of fresh and frozen-warmed single blastocyst transfer: a 5-year single-center experience. J Assist Reprod Genet. 2022 Jan;39(1):201-209. doi: 10.1007/s10815-021-02362-3. Epub 2021 Nov 26. PMID 34837160